CLINICAL TRIAL: NCT06161194
Title: Efficacy of Real-time Feedback Exercise Therapy in Patients Following Total Hip Arthroplasty: a Pilot Cluster-randomized Controlled Trial
Brief Title: Efficacy of Real-time Feedback Exercise Therapy in Patients Following Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaus Widhalm (Other)
Collaborators: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Sponsor-Investigator, Klaus Widhalm, Head of study, FH Campus Wien, University of Applied Sciences
Organization: FH Campus Wien, University of Applied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP_SETT_RCT-THA
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hip Replacement
Keywords: hip replacement; exercise therapy; real-time feedback; movement analysis

STUDY DESIGN:
Intervention Model Description: cluster-randomized, two-arm parallel-group controlled trial
Masking Description: Participants will be randomly assigned to IG or CG after baseline assessment. Due to the nature of the studied conditions, it will not be possible to blind researchers or participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (IG) (Experimental): IG will perform the home-exercise program supported by the digital real-time exercise feedback prototype for digitally guided training.
  Interventions: Other: Supervised group exercise therapy
- Control Group (CG) (Active Comparator): The CG will perform a usual care home-exercise by means of printed hand-outs describing each exercise.
  Interventions: Other: Supervised group exercise therapy

INTERVENTIONS:
Other: Supervised group exercise therapy — Participants will participate in a 90 minutes supervised group exercise therapy program 2 times a week for 8 consecutive weeks.

SUMMARY:
This pilot cluster-randomized, two-arm parallel-group controlled trial, aims at enhancing the understanding of the effects of real-time feedback on functional deficits as knee valgus thrust, pelvic drop, and lateral trunk lean after total hip arthroplasty. Biomechanical and patient-reported outcomes will be assessed after a total hip arthroplasty as well as at three and six months follow-ups. The primary research question is, whether digital real-time feedback supported home-exercising improves the control of the frontal knee range of motion, pelvic obliquity, and lateral trunk lean, superior to exercising supported by written instructions as comparator. The secondary aspect focuses on potential differences between groups concerning aspects of quality of life, function, and physical activity. Tertiary functional outcomes between groups will be compared for reasons of quantification movement quality.

ELIGIBILITY:
Inclusion Criteria:

* age from 50-75 years
* body mass index from 18.5 to 29.99 kg/m²
* able to walk without walking aids at baseline assessment
* scheduled for elective unilateral total hip arthroplasty surgery
* willing to comply with all study related procedures and provide informed consent

Exclusion Criteria:

* symptoms of delayed healing concerning the implant
* cardio-respiratory symptoms limiting exercise therapy (for example severe heart disease)
* symptoms of musculoskeletal or cardio-respiratory overload
* neuro-motor diseases (for example previous Stroke, Multiple Sclerosis, Morbus Parkinson Disease)
* other reasons which would lead to obvious limitations concerning their participation in the intervention (for example severe contralateral osteoarthritis (OA), lower extremity fractures within previous 12 months, other elective lower extremity surgery within 6 months, inadequacy in German concerning questionnaires and exercise instructions, mentally unable to participate)
* non-adherence (see definition under "therapeutic adherence").

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Frontal knee angle range of motion Pelvic obliquity angle range of motion Frontal trunk angle range of motion | Baseline 4 weeks post-surgery; 3-months post-surgery; 6-months post-surgery
  Above listed angles derived from assessed Activities of Daily Living (ADL) tasks

SECONDARY OUTCOMES:
Harris Hip Score (HHS) Hip Osteoarthritis Outcome Score (HOOS) Short-Form-Health Survey (SF12) International Physical Activity Questionnaire - short form (IPAQ) if applicable: Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline 4 weeks post-surgery; 3-months post-surgery; 6-months post-surgery

OTHER OUTCOMES:
3D-movement-analysis parameters (kinematic, kinetic, spatio-temporal) | Baseline 4 weeks post-surgery; 3-months post-surgery; 6-months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Widhalm, Study Director — FH Campus Wien, University of Applied Sciences
Locations (1):
- Orthopaedic Hospital Vienna Speising, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The study protocol including the statistic analysis plan will be submitted for publication in Trials Journal at begin of 2024.
  The final results will be submitted for publication to a relevant journal by the end of 2025.
Access Criteria: Open Access publication

REFERENCES:
- [Derived] Widhalm K, Maul L, Durstberger S, Putz P, Leder-Berg S, Kainz H, Augat P. Efficacy of Real-Time Feedback Exercise Therapy in Patients Following Total Hip Arthroplasty: Protocol for a Pilot Cluster-Randomized Controlled Trial. JMIR Res Protoc. 2024 Aug 20;13:e59755. doi: 10.2196/59755. PMID 39163589